CLINICAL TRIAL: NCT03900403
Title: The Influence of Daily Walnut Intake on Vascular Function and Associated Changes in Lipid Mediators and Primary Metabolites.
Brief Title: Influence of Walnut Intake on Vascular Function and Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1313232
Record Dates: First submitted 2019-03-31; First posted 2019-04-03 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Overweight and Obesity; Endothelial Dysfunction; Cardiovascular Risk Factor
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Open-arm study, comparing the effects of 12 weeks of 40g of walnut intake to 6 weeks of the study participant's habitual diet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Habitual Intake (No Intervention): This will be the comparative arm, of 6 weeks before and after the study participant is on their habitual diet
- Walnut Intake (Experimental): Experimental Arm of 12 weeks of Walnut Intake, with study visits at baseline (prior to walnut intake) and after 6 and 12 weeks of 40g of Walnut Intake.
  Interventions: Other: Walnut Intake

INTERVENTIONS:
Other: Walnut Intake — 40g of daily walnut intake for 12 weeks
  Arms: Walnut Intake

SUMMARY:
This study seeks to confirm and extend previous finding that four weeks of daily intake of 40 g of walnuts improve microvascular function, increasing the reactive hyperemia index (RHI), effects which were greatest in individuals with the worst initial RHI and correlating to circulating levels of vasoactive plasma epoxides. The current trial will enroll postmenopausal women who are at risk for cardiovascular disease due to their menopausal status and increased central adiposity. The initial trial focused on non-esterified (i.e. plasma) derived oxylipins, but substantial and unique changes were also observed in the esterified lipoprotein pool. The current study will add the esterified lipoprotein pool, important, as the mechanisms by which walnut intake influences endothelial function are currently undefined, but may include lipoprotein induced modulation of vascular hemostasis. As a secondary objective, primary metabolism and urolithin metabotype will be analyzed as a way to capture the influence of potential differences in habitual diet and metabolism on physiologic response. Therefore, this study will combine measures of cardiovascular physiology, metabolomics, and walnut-derived metabolite analyses to assess the 12 week influence of 40 g of daily walnut intake on the health of overweight and obese postmenopausal women.

DETAILED DESCRIPTION:
A dietary intervention trial will be conducted to achieve the following objectives and outcomes:

Objective 1: Determine the 12 week change in bioactive lipid mediators, and their relationship to vascular function and platelet reactivity in overweight or obese postmenopausal women with walnut incorporation into their habitual diet.

Objective 2: Assess the contribution of metabolic phenotype on the variance in biomarker response that includes both primary metabolism and urolithin metabotype.

Expected Outcomes: Forty g of daily walnut intake for six- and 12- weeks is predicted to positively impact the production of bioactive lipid mediators known to favorably regulate cardiovascular and inflammatory signaling. AA derived oxylipins produced from COX, LOX, and CYP epoxygenases are known as regulators of inflammation, platelet activation and vascular function. Therefore, understanding how certain foods such as walnuts can change the relative ratio of PUFA substrates (i.e., AA, ALA, LA, EPA and DHA), and their subsequent bioactive species produced through these enzyme pathways is necessary for the refinement of dietary recommendations with regard to specific foods and dietary patterns aimed at reducing the risk of chronic disease. Although a positive outcome is predicted, there may be substantial variability in response. To explore potential genetic and dietary factors that may contribute to the variability in response to the above functional markers, primary metabolism and urolithin metabotype will be assessed.

Objective 3: Assess the influence of 12 weeks of walnut intake on facial wrinkles in postmenopausal women.

Expected Outcome: Tweleve weeks of 40 g of walnut intake will improve facial wrinkles and erythema in the study population, and the improvements will be related to changes in metabotype.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female: 45-65 years
* Women: lack of menses for at least two years.
* Subject is willing and able to comply with the study protocols.
* Subject is willing to participate in all study procedures
* BMI 25.0 - 35 kg/m2

Exclusion Criteria:

* BMI ≥ 35 kg/m2
* Visit 1 Reactive Hyperemia Index (RHI; EndoPAT 2000) ≥ 2.4
* Dislike or allergy for walnuts or walnut products
* Self-reported use of daily anticoagulation agents including aspirin, NSAIDs
* Vegan, Vegetarians, food faddists or those consuming a non-traditional diet
* Fruit consumption ≥ 3 cups/day
* Regular consumption of nuts (2-3 servings/week)
* Vegetable consumption ≥ 4 cups/day for females
* Coffee/tea ≥ 3 cups/day
* Dark chocolate ≥ 3 oz/day
* Self-reported restriction of physical activity due to a chronic health condition
* Self-reported chronic/routine high intensity exercise
* Self-reported diabetes
* Blood pressure ≥ 140/90 mm Hg
* Self-reported renal or liver disease
* Self-reported heart disease, which includes cardiovascular events and stroke
* Peripheral artery disease, Raynaud's syndrome or disease
* Inability to properly place or wear the PAT probes or abnormal measurements on pre-screening PAT
* Abnormal Metabolic or CBC panels (laboratory values outside the reference range) if determined to be clinically significant by the study physician.
* Self-reported cancer within past 5 years
* Self-reported malabsorption
* Currently taking prescription drugs or supplements.
* Supplement use other than a general formula of vitamins and minerals that meet the RDA
* Not willing to stop any supplement use, including herbal, plant or botanical, fish oil, oil supplements a month prior to study enrollment.
* Indications of substance or alcohol abuse within the last 3 years
* Cannabis use
* Screening LDL ≥ 190 mg/dl for those who have 0-1 major risk factors apart from LDL cholesterol (i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL]. (using NCEP calculator http://cvdrisk.nhlbi.nih.gov/calculator.asp)
* Screening LDL ≥ 160 mg/dl for those who have 2 major risk factors apart from LDL cholesterol [i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL]. (using NCEP calculator http://cvdrisk.nhlbi.nih.gov/calculator.asp);
* Screening LDL ≥ 130 mg/dl for those who have 2 major risk factors apart from LDL cholesterol [i.e. family history of premature coronary artery disease (male first degree relative < 55 years; CHD in female first degree relative < 65 years), cigarette smoker, HDL-C ≤ 40 mg/dL], and a Framingham 10-year Risk Score 10-20% (using NCEP calculator http://cvdrisk.nhlbi.nih.gov/calculator.asp).
* Current enrollee in a clinical research study.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
Reactive Hyperemia Index (RHI) | 18 weeks
  Digital microvascular function as measured by the EndoPAT2000
Framingham Reactive Hyperemia Index (fRHI) | 18 weeks
  Digital microvascular function as measured by the EndoPAT2000

SECONDARY OUTCOMES:
Collagen-Induced Platelet Aggregation | 18 weeks
  Optical platelet aggregometry
ADP-Induced Platelet Aggregation | 18 weeks
  Optical platelet aggregometry
Plasma Fatty Acids | 18 weeks
  Circulating levels of non-esterified fatty acids
Plasma Oxylipins | 18 weeks
  Circulating levels of non-esterified oxylipins
Esterified Oxylipins | 18 weeks
  Lipoprotein esterified oxylipins
Esterified Fatty Acids | 18 weeks
  Lipoprotein esterified fatty acids
Urolithin Metabolites | 18 weeks
  Conjugated and unconjugated urolithins
Ellagitannin Metabolites | 18 weeks
  Conjugated and unconjugated Ellagitanin-derived metabolites
Total Nitrate and Nitrite | 18 weeks
  Total nitrate derived from the diet
Nitric Oxide metabolites (RNOX) | 18 weeks
  Nitric oxide metabolites produced from the intervention

OTHER OUTCOMES:
Blood Pressure | 18 weeks
  Office blood pressure
Complete Metabolic Panel | 18 weeks
  Will include liver enzymes and glucose
Complete Blood Cell Count | 18 weeks
  w Will include total platelet number and mean platelet volume
Lipid Panel | 18 weeks
  Will assess fasting cholesterol and triglyceride levels
Skin Health | 18 weeks
  Will assess fine facial wrinkles and redness

CONTACTS AND LOCATIONS:
Overall Officials: Roberta R Holt, PhD, Principal Investigator — University of California, Davis
Locations (1):
- Department of Nutrition, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/walnut-study-411535/